CLINICAL TRIAL: NCT03499197
Title: Morphological and Functional Changes After Heart Transplantation - Role of Noninvasive Imaging in the Early Detection of Cardiac Allograft Rejection and Vasculopathy
Brief Title: Heart TIMING - Heart Transplantation IMagING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: National Research, Development and Innovation Fund of Hungary, Project no. NVKP_16-1-2016-0017 (Unknown)
Responsible Party: Principal Investigator, Hajnalka Vágó MD PhD, MD PhD, Associate Professor, Semmelweis University Heart and Vascular Center
Other Study IDs: Heart TIMING 001
Record Dates: First submitted 2018-04-11; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Heart Transplant Failure and Rejection; Magnetic Resonance Imaging
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cardiac magnetic resonance imaging — Detailed and regular CMR examination (LGE, stress perfusion, T1, T2 mapping)

SUMMARY:
The cardiac allograft rejection (CAR) and cardiac allograft vasculopathy (CAV) significantly affect the prognosis of patients after heart transplantation. The aim of the present study is to investigate and differentiate the adaptive and pathological cardiovascular changes after heart transplantation using different modalities. The investigator's main purpose is to define the role of the cardiovascular imaging methods and biomarkers in the early diagnosis of CAR and CAV.

DETAILED DESCRIPTION:
1. 12-lead ECG - Resting standard 12-lead digital ECG will be recorded. Extended analysis will be performed according to the latest recommendations.
2. Holter ECG - 24 hour Holter ECG will be recorded. Extended Holter ECG analysis will be performed.
3. Life quality questionnaire, patient history - Detailed questionnaire about personal and family history, general symptoms and life quality.
4. Laboratory biochemical examination - Besides the regular routine laboratory parameters, several specific parameters are planned to be measured, such as cardiac biomarkers.
5. Endomyocardial biopsy
6. Detailed transthoracic echocardiography including strain analysis and 3D measurement
7. Detailed cardiac magnetic resonance (CMR) examination
8. Coronary imaging - invasive coronarography and intravascular ultrasound (IVUS) and/or optical coherence tomography (OCT)
9. Invasive pressure measurement - Measurement of coronary flow reserve (CFR) and microcirculation resistance index (IMR)

ELIGIBILITY:
Inclusion Criteria:

* First heart transplantation

Exclusion Criteria:

* Cardiogenic shock on/after day 28 after heart transplantation
* Lack of consent
* Lack of cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent first cardiac transplantation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Coronary allograft vasculopathy | 5 years
  Coronary allograft vasculopathy confirmed based on IVUS/OCT
Coronary allograft rejection | 5 years
  Coronary allograft rejection confirmed based on endomyocardial biopsy/clinical parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Heart and Vascular Center, Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided